CLINICAL TRIAL: NCT06581705
Title: The C-MAC Video Laryngoscope Helps Presbyopic Anesthetists to Overcome Difficulty in Neonatal and Infantile Intubation. A Randomized Controlled Trial
Brief Title: The C-MAC Video Laryngoscope Helps Presbyopic Anesthetists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: The C-MAC Video
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: (video laryngoscope Group) (Active Comparator): About 50 anesthetists in charge must be older than 40 years; each anesthetist had to manage at least 10 patients from both groups received endotracheal intubation (ETI) using the SL and VL group had intubated using the C-MAC® (Karl Storz, Germany) VL with the standard Miller blade and flexible Stylet (2 mm PORTEX® stylet; Smiths Medical International Ltd., UK) to strengthen the endotracheal tube (ETT) and adjust its curvature as C-shaped. The study outcomes included the frequency of successful intubation within 30 s (30-s SR) and the number of intubation attempts. .
  Interventions: Procedure: Video Laryngoscope
- Group B: (Standard laryngoscope Group) (Active Comparator): About 50 anesthetists in charge must be older than 40 years; each anesthetist had to manage at least 10 patients from both groups received endotracheal intubation (ETI) using the SL and VL group had intubated using the C-MAC® (Karl Storz, Germany) VL with the standard Miller blade and flexible Stylet (2 mm PORTEX® stylet; Smiths Medical International Ltd., UK) to strengthen the endotracheal tube (ETT) and adjust its curvature as C-shaped. The study outcomes included the frequency of successful intubation within 30 s (30-s SR) and the number of intubation attempts. .
  Interventions: Procedure: Video Laryngoscope

INTERVENTIONS:
Procedure: Video Laryngoscope — Evaluation of the success rates (SR) of anesthetists aged ≥45 years for intubating neonates and infants using the C-MAC videolaryngoscope (VL) in comparison to the use of the standard laryngoscope (SL).

SUMMARY:
Endotracheal intubation is the de facto gold standard for airway management especially in neonatal and pediatric anesthesia .

An efficient neonatal airway management is challenging even in the most experienced hands and the prevalence of difficult intubation in pediatric anesthesia varied greatly on a wide range.

DETAILED DESCRIPTION:
Neonatal intubation is a life-saving procedure, which requires skilled operator but still may cause direct tissue trauma and precipitate adverse reactions. However, intubation with videolaryngoscope (VL) requires less force than with a direct laryngoscope to minimize the possibility of these adverse events.

The recent Brazilian recommendations for management of pediatrics difficult airways included proper assessment, preparation, positioning, pre-oxygenation, minimizing trauma, maintenance of arterial oxygenation and the implementation of the advanced tools as VL, flexible intubating bronchoscopy, and supraglottic devices.

The recent British recommendations also advised for the use VL with an age-adapted standard blade as first choice for tracheal intubation and the use of a stylet to reinforce and preshape tracheal tubes in case of the use of hyperangulated VL blades .

Considering the recent interest in assessing the performance of various VLs in pediatric anesthesia, the C-MAC® (Karl Storz, Germany) VL with standard Miller blade sizes #0 and #1, is a widely used in neonates and infants for its provision of superior-quality glottis view in comparison to the McGrathTM MAC size #1 blade and direct laryngoscopy.

Presbyopia is defined as disordered eye adjustment function and affects middle aged people leading to difficult viewing close objects and is corrected with magnifying lens.

Earlier studies documented that presbyopic aged anesthetists find difficulty when trying to view a patient's larynx at a close distance and this difficulty is surely magnified on dealing with intubation of neonates and children

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients whom scheduled for surgical procedures under general inhalation anesthesia

Exclusion Criteria:

* Patients older than 12 months
* patients with Mallampati score of 3 or 4,
* patients had abnormal airway and obstructive sleep apnea,
* manifestations of upper respiratory tract infection or uncompensated cardiopulmonary diseases
* patients with ASA grade >III were excluded from this study.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
the frequency of successful intubation | 30 seconds
  The frequency of the need for external laryngeal manipulation, head extension, or stylet curvature change to achieve intubation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M.Elnagar, M.D, Principal Investigator — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Abdalla AE, Eissa MM, Elbasyouny MR, Zomra MR, Elnaggar AM, Elsayed MM. The C-MAC video laryngoscope helps presbyopic anesthetists to overcome difficulty in neonatal and infantile intubation: a randomized controlled trial. BMC Anesthesiol. 2025 Jan 10;25(1):24. doi: 10.1186/s12871-024-02841-x. PMID 39794694